CLINICAL TRIAL: NCT04012138
Title: InSaKa Trial: Insulin Dextrose Infusion Versus Nebulized Salbutamol Versus Combination of Salbutamol and Insulin Dextrose in Acute Hyperkalemia: a Randomized Clinical Trial
Brief Title: Insulin Dextrose Infusion vs Nebulized Salbutamol vs Combination of Salbutamol and Insulin Dextrose in Acute Hyperkalemia
Acronym: InSaKa
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC19_0048
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hyperkalemia
Keywords: hyperkaliema; insulin; salbutamol
MeSH Terms: conditions — Hyperkalemia; Insulin Resistance | interventions — Albuterol; Insulin Aspart; Insulin

STUDY DESIGN:
Intervention Model Description: InSaKa trial is a therapeutic, controlled, open label, with parallel groups of treatment in a 1:1:1 ratio, multi-centre, national and randomized clinical trial to compare insulin/dextrose intravenous infusion, nebulized salbutamol or combination of salbutamol and insulin/dextrose to reduce serum potassium levels at 60 minutes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Salbutamol (Experimental): Patients in this experimental group will receive : 10 mg of salbutamol nebulized in 30 minutes (with oxygen 8 liters per minute or with air);
  Interventions: Drug: Salbutamol
- Insuline + dextrose (Active Comparator): Patients in the experimental group will receive : 10 units of regular insulin (rapid-acting, insuline asparte, intravenous injection) as an intravenous bolus with 500 ml of 10% dextrose in water administered over a 30-minute period
  Interventions: Drug: Insulin Aspart
- Insuline + Dextrose + Salbutamol (Experimental): Patients in the experimental group will receive either:
  1. 10 mg of salbutamol nebulized in 30 minutes (with oxygen 8 liters per minute or with air); OR
  2. 10 units of regular insulin (rapid-acting, insuline asparte, intravenous injection) as an intravenous bolus with 500 ml of 10% dextrose in water administered over a 30-minute period plus 10 mg of salbutamol nebulized in 30 minutes (with oxygen 8 liters per minute or with air). The nurse will start by giving the 10 units of insulin and the dextrose, and then, immediately, she will start the nebulization of salbutamol.
  Interventions: Drug: Salbutamol; Drug: Insulin Aspart

INTERVENTIONS:
Drug: Salbutamol — 10 mg of salbutamol nebulized in 30 minutes (with oxygen 8 liters per minute or with air) 10 units of regular insulin (rapid-acting, insuline asparte, intravenous injection) as an intravenous bolus with 500 ml of 10% dextrose in water administered over a 30-minute period.
  Other Names: Salbutamol and Hyperkaliemia
  Arms: Insuline + Dextrose + Salbutamol; Salbutamol
Drug: Insulin Aspart — Patients in the experimental group will receive either:
  1. 10 mg of salbutamol nebulized in 30 minutes (with oxygen 8 liters per minute or with air); OR
  2. 10 units of regular insulin (rapid-acting, insuline asparte, intravenous injection) as an intravenous bolus with 500 ml of 10% dextrose in water administered over a 30-minute period plus 10 mg of salbutamol nebulized in 30 minutes (with oxygen 8 liters per minute or with air). The nurse will start by giving the 10 units of insulin and the dextrose, and then, immediately, she will start the nebulization of salbutamol.
  Other Names: Insulin and Hyperkaliemia
  Arms: Insuline + Dextrose + Salbutamol; Insuline + dextrose

SUMMARY:
Hyperkalemia is a common electrolyte disorder, especially among patients with chronic kidney disease, diabetes mellitus, or heart failure. Globally, the reported incidence of hyperkalemia varies from 1.1 to 10 per 100 hospitalizations, depending on the patient cohort and comorbidities. Hyperkalemia is a potentially life-threatening electrolyte disturbance that can be fatal if left untreated. Several studies have established the association between hyperkalemia and all-cause mortality. Because of the deleterious cardiac effects of hyperkalemia, its management is an emergency intervention. However, robust evidence is lacking to guide the emergency management of patients with hyperkalemia. Emergency treatment approaches are largely based on small studies, anecdotal experience, and traditionally accepted practice patterns within institutions. Therefore, a rigorous evaluation of the first-line treatments of hyperkalemia in emergency departments is needed and a large scale randomized clinical trial is warranted before robust recommendations for clinical practice can be made. Our clinical trial will improve the safety of patients with acute hyperkalemia and will help clinicians in their day by day practice to choose the treatment that significantly reduces morbidity and mortality during acute hyperkalemia management. Our results will be delivered in a timely fashion, owing to the high prevalence of hyperkalemia in the emergency department setting and to the commitment of the INI-CRCT network of Excellence, along with ED specialists used to work jointly.

the primary objective of our trial is to compare insulin/dextrose intravenous infusion, nebulized salbutamol or combination of nebulized salbutamol and insulin/dextrose intravenous infusion to reduce serum potassium concentration at 60 minutes, as first-line treatment, in emergency departments.

DETAILED DESCRIPTION:
InSaKa trial is a therapeutic, controlled, open label, with parallel groups of treatment in a 1:1:1 ratio, multi-centre, national and randomized clinical trial to compare insulin/dextrose intravenous infusion, nebulized salbutamol or combination of salbutamol and insulin/dextrose to reduce serum potassium levels at 60 minutes. Eligible patients will be recruited in the emergency department and included in the study after testing for inclusion and non-inclusion criteria. Patients will be eligible for the randomization if they had a serum potassium concentration superior or equal to 6 mmol per liter. Randomization, which will be performed centrally, will be stratified 1) according to the serum potassium level at baseline of the initial treatment phase (6 to < 6.5 mmol per liter [moderate hyperkalemia] AND superior or equal to 6.5 mmol per liter [severe hyperkalemia]), and 2) according to the prescription or not of intravenous diuretics during the 6 previous hours. The protocol will be approved by the ethical committee (random allocation) of the IRB. All patients will provide written informed consent and the study will be performed in accordance with the International Conference on Harmonization Guidelines for Good Clinical Practice. All electrocardiograms will be read at a core electrocardiographic laboratory. At the time of screening, patients who meet all the inclusion and do not have non-inclusion criteria will be assigned to one of the 3 groups of treatment. The serum potassium will be then measured at 60 minutes. If the patient still has hyperkalemia at 60 minutes, the patient will be re-administered a treatment, left at the discretion of the physician in charge. This treatment might include insulin/dextrose intravenous infusion, nebulized salbutamol, the combination of nebulized salbutamol and insulin/dextrose intravenous infusion, bicarbonate, diuretics or dialysis. Especially, bicarbonate should be prescribed in case of metabolic acidosis or hypovolemic shock, and diuretics in case of acute heart failure. Importantly, if the patient has a major cardiovascular event before 60 minutes, all these treatments might be prescribed at the discretion of the physician in charge, if the clinical situation requires one or more of these therapeutic options, and based on up-to-date clinical practice guidelines and recommendations. Serum potassium levels will be measured at local laboratories at baseline and 60, 180 minutes and 24 hours. They will perform a visual inspection and a validated semi-quantitative test on each blood sample as an assessment for hemolysis. An independent adjudication committee will adjudicate all major cardiovascular events. The trial will be monitored by a Data Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient admitted to the emergency department,
* Patient with local laboratory serum potassium level superior or equal to 5,5 mmol/l,
* Patient who provide written informed consent prior to participation in the study

Exclusion Criteria:

* Hemolysis or thrombocytosis > 106/mm3 or hyperleukocytosis > 105/mm3 on the first blood sample suspecting a pseudohyperkalemia,
* Diabetic ketoacidosis or hyperosmolar hyperglycemic syndrome,
* Pregnant or lactating woman, women with childbearing potential who didn't have effective contraception*,
* Patient expected to require emergency intubation and ventilation,
* Patient expected to require dialysis, diuretics or bicarbonate within the first 60 minutes,
* Patient with heart rhythm disorders or high grade atrioventricular bloc who require urgent medication as soon as admission or serum potassium level result,
* Hypersensitivity to the tested active substance or excipients,
* Acute coronary syndrome,
* Patient not affiliated to a health insurance plan,
* Patient under guardianship, curatorship or safeguard of justice.

  * The contraceptives considered as highly effective and acceptable by CTFG recommendations will be considered effective under this protocol. The list of contraceptives considered as highly effective and acceptable by CTFG recommendations is detailed in Appendix 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Mean change in the absolute serum potassium level from baseline to 60 minutes | 60 minutes
  The primary outcome of our trial will be mean change in the absolute serum potassium level from baseline to 60 minutes (measured in mmol/l), and will be aggregated using median and interquartile.

SECONDARY OUTCOMES:
Mean change in the serum potassium level from baseline to 180 minutes and 24 hours | 180 minutes and 24 hours
Proportion of patients who had a serum potassium level of 4 mmol/l to less than 4.9 mmol/l at 60, 180 minutes and 24 hours | 60 minutes, 180 minutes and 24 hours
Proportion of patients who require re-treatment or dialysis at 60, 180 minutes and 24 hours | 60 minutes, 180 minutes and 24 hours
Proportion of patients with adverse effects at 60 and 180 minutes | 60 minutes and 180 minutes
  Proportion of patients with adverse effects at 60 and 180 minutes :
  1. Hypokalemia (serum potassium level <3.5 mmol/l and <4 mmol/l)
  2. Hypomagnesemia (serum magnesium level of less than 0.58 mmol per liter)
  3. Hypoglycemia (serum glucose level < 4.0 mmol/l)
  4. Hyperglycemia (serum glucose level > 10.0 mmol/l)
  5. Gastrointestinal disorders:
  i. Diarrhea ii. Nausea iii. Vomiting f. Tachycardia (> 130/min) g. Tremor
Proportion of patients with heart rhythm disorders or high grade atrioventricular bloc that required urgent medication during the first 180 minutes | 180 minutes
Proportion of patients with electrocardiographic abnormalities, at 60, 180 minutes and 24 hours | 60 minutes 180 minutes and 24 hours
  Proportion of patients with electrocardiographic abnormalities, at 60, 180 minutes and 24 hours , including:
  1. Auricular extrasystoles
  2. Ventricular extrasystoles
  3. Atrioventricular block
  4. QRS Interval Prolongation (> 120 ms)
  5. QT interval prolongation (> 500 ms)
Proportion of major cardiovascular events at 60, 180 minutes and 24 hours | 60minutes 180 minutes and 24 hours
  Proportion of major cardiovascular events at 60, 180 minutes and 24 hours :
  1. cardiac arrest
  2. stroke
  3. acute heart failure
  4. complete atrioventricular block with ventricular rate under 30 bpm
  5. ventricular fibrillation
  6. ventricular tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Julie CONTENTI, Principal Investigator — Nice University Hopsital; Pierre-Clément THIEBAUD, Principal Investigator — Saint Antoine University Hospital; Maxime MAIGNAN, Principal Investigator — University Hospital, Grenoble; Jeannot SCHMIDT, Principal Investigator — University Hospital, Clermont-Ferrand; Meïssa KARE, Principal Investigator — Agen Hospital; Tahar CHOUIHED, Principal Investigator — Central Hospital, Nancy, France; Anne-Laure FERAL-PIERSSENS, Principal Investigator — Avicenne University Hospital; Florent MAILLET, Principal Investigator — Louis Mourier Hospital; Quentin DELANNOY, Principal Investigator — La Pitié Salpetrière University Hospital; Nicolas MARJANOVIC, Principal Investigator — Poitiers University Hospital; delphine DOUILLET, Principal Investigator — Angers University Hospital; Paul-Louis MARTIN, Principal Investigator — Tours University Hospital; Pierrick LE BORGNE, Principal Investigator — University Hospital, Strasbourg, France; Xavier EYER, Principal Investigator — Lariboisière Hospital; Nicolas PESCHANSKI, Principal Investigator — Rennes University Hospital
Locations (16):
- France (16):
  - Agen Hospital, Agen
  - Angers University Hospital, Angers
  - Avicenne University Hospital, Bobigny
  - University Hospital, Clermont-Ferrand, Clermont-Ferrand
  - Louis Mourier Hospital, Colombes
  - University Hospital, Grenoble, Grenoble
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - La Pitié Salpêtrière University Hospital, Paris
  - Lariboisiere Hospital, Paris
  - Saint Antoine University Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Strasbourg University Hospital, Strasbourg
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: Yes
Trial data are not publicly available owing to data privacy, but access to the anonymised dataset can be obtained from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: the dataset can be obtained from the corresponding author on reasonable request

REFERENCES:
- [Derived] Montassier E, Lemoine L, Hardouin JB, Rossignol P, Legrand M. Insulin glucose infusion versus nebulised salbutamol versus combination of salbutamol and insulin glucose in acute hyperkalaemia in the emergency room: protocol for a randomised, multicentre, controlled study (INSAKA). BMJ Open. 2020 Aug 26;10(8):e039277. doi: 10.1136/bmjopen-2020-039277. PMID 32847923